CLINICAL TRIAL: NCT06884059
Title: Impact of Time-Restricted Eating (TRE) on Kidney Health (The TREK Study)
Brief Title: Time Restricted Eating in Patients With Microalbuminuria
Acronym: TREK
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Salk Institute for Biological Studies (Other)
Responsible Party: Principal Investigator, Pam Taub, MD, Pam Taub, MD, Professor of Medicine, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 810456
Record Dates: First submitted 2025-03-05; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-01

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Time Restricted Eating; Microalbuminuria
Keywords: Microalbuminuria; Time Restricted Eating; Urine Albumin-to-Creatinine Ratio; Type 2 Diabetes; uACR; Fasting
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Intermittent Fasting; Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Time Restricted Eating (TRE) Group (Experimental): Participants will limit the number of hours they eat in a dat to an 8-10 window and will also receive the standard heath and nutritional wellness guidelines. They will also be required to log food entries through the use of a smartphone app. Patients will also be required to wear a continuous glucose monitor (CGM) for the first and last two weeks of the 14 trial.
  Interventions: Behavioral: Time Restricted Eating

INTERVENTIONS:
Behavioral: Time Restricted Eating — Participants in the TRE group with continue to follow their physicians treatment plan for type II diabetes mellitus and consume all of their food within an 8-10 hour eating window.

SUMMARY:
This is a clinical trial to assess how time-restricted eating (TRE) may improve kidney health and filtration patients with type 2 diabetes and increased protein content in their urine. All participants will be participating in TRE in which they follow a consistent 8-10 hour eating window everyday.

DETAILED DESCRIPTION:
The proposed study aims to address the unmet medical need of treating microalbuminuria, particularly in patients with diabetes, through a prospective single-arm intervention lasting twelve weeks. Microalbuminuria, indicative of abnormal glomerular capillary permeability, serves as an early marker for renal impairment and heightened cardiovascular risk. The study hypothesizes that adherence to time-restricted eating (TRE) over the intervention period will significantly reduce microalbuminuria levels, as assessed by the urine albumin-to-creatinine ratio (uACR). Unlike other methods, uACR provides an estimation of 24-hour urine albumin excretion and is unaffected by variations in urine concentration, eliminating the need for timed specimens or 24-hour collections. If successful, this study could highlight the potential of TRE as a non-invasive and accessible dietary intervention for managing microalbuminuria and related conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years old
2. Participants with T2DM with A1c between 6.5 and 9.0 % and on stable doses of medications who are weight-bearing and self-ambulatory.
3. uACR ( urine albumin creatinine ratio) results ≥ 30 - 300 mg.
4. Willingness to use smartphone for research procedures (Apple iOS or Android OS)
5. Baseline eating period ≥12 hours/day and sufficient logging on the mCC app.
6. Person of childbearing potential will be given a pregnancy test on study enrollment and asked to use contraception throughout the study.
7. Post-menopausal and individuals on hormone replacement therapy will be included.
8. Estimated Glomerular Filtration Rate (EGFR) > 45
9. If participants are on cardiovascular medications (HMG CoA reductase inhibitors (statins), other lipid-modifying drugs, anti-hypertensives) no dose adjustments will be allowed during the study period
10. Participants on stable doses (consistent dose for ≥3 months) of GLP-1 receptor agonists will be included.

Exclusion Criteria:

1. Participants with Type1DM and T2DM who are taking insulin, sulfonylureas, or have an HbA1c > 9 %.
2. Estimated Glomerular Filtration Rate (EGFR) < 45
3. Systolic BP greater than 160 mmHg and/or Diastolic BP greater than 110 mmHg (with or without treatment/medication)
4. LDL cholesterol greater than 200 mg/dL
5. Triglycerides greater than 500 mg/dL
6. Active tobacco or illicit drug use
7. Pregnant or breastfeeding individuals.
8. Currently enrolled in a weight-loss or weight-management program,
9. Currently on a special or prescribed diet for other reasons (e.g., Celiac disease),
10. On recently prescribed medication that is meant for weight loss, or has known effect on appetite suppression ( patient on stable dose for 3 months can be enrolled ).
11. History of eating disorder(s).
12. History of surgical intervention for weight management (e) active eating disorder.
13. Chronic kidney disease with an eGFR calculated based on the Modification of Diet in Renal Disease (MDRD) equation <50mL/min/1.73m2
14. Treatment for active inflammatory and/or rheumatologic disease and cancer.
15. A major adverse cardiovascular event within the past 6 months such as acute coronary syndrome (ACS), percutaneous coronary intervention, coronary artery bypass graft surgery, hospitalization for congestive heart failure, stroke/transient ischemic attack (TIA).
16. History of Uncontrolled arrhythmia (i.e., rate-controlled atrial fibrillation/atrial flutter are not exclusion criteria) 18. Liver cirrhosis and/or significant alterations in liver function
17. History of (a) thyroid disease requiring dose titration of thyroid replacement medication(s) within the past 3 months (i.e., hypothyroidism on a stable dose of thyroid replacement therapy is not an exclusion), Shift workers with variable (e.g., nocturnal) hours.
18. Caregivers for dependents requiring frequent nocturnal care/sleep interruptions.
19. More than one trip planned to travel to a time zone with greater than a 3-hour difference during study period.
20. History of major adverse cardiovascular events within the past 1 year (acute coronary syndrome (ACS), percutaneous coronary intervention, coronary artery bypass graft surgery, hospitalization for congestive heart failure, stroke/transient ischemic attack (TIA)).
21. History of thyroid disease requiring dose titration of thyroid replacement medication(s) within the past 3 months (i.e., hypothyroidism on a stable dose of thyroid replacement therapy is not an exclusion).
22. History of adrenal disease.
23. History of malignancy undergoing active treatment, except non-melanoma skin cancer.
24. Known history of type I diabetes.
25. History of stage 4 or 5 chronic kidney disease or requiring dialysis.
26. History of HIV/AIDS.
27. Uncontrolled psychiatric disorder (including history of hospitalization for psychiatric illness).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Urine albumin-to-creatinine ratio (uACR) | Baseline and 3 months
  Change in uACR (mg/g) assessed via urine sample

SECONDARY OUTCOMES:
Glycemic regulation assessed by Continuous Glucose Monitor (CGM) | Baseline and 3 months
  Change in glycemic regulation as assessed by CGM from interstitial glucose with various outcomes measured.
Fasting glucose levels (mg/dL) | Baseline and 3 months
  Change in glycemic regulation as assessed fasting plasma glucose (mg/dL).
Glycemic regulation assessed by HbA1c | Baseline and 3 months
  Change in blood glucose assessed via hemoglobin A1c.
Blood pressure | Baseline and 3 months
  Change in blood pressure assessed by sphygmomanometer.
LDL-Cholesterol | Baseline and 3 months
  Changes in atherogenic lipids assessed via LDL-Cholesterol.
Non-HDL Cholesterol (nmol/mol) | Baseline and 3 months
  Changes in atherogenic lipids assessed via LDL-Cholesterol.
Triglycerides (mg/dL) | Baseline and 3 months
  Changes in atherogenic lipids assessed via Triglycerides (mg/dL).
Quality of life Assessment via Short Form-36 Questionnaire (SF-36) | Baseline and 3 months
  Changes in quality of life will be assessed using the SF-36 questionnaire, with scores ranging from 0 to 100, where higher scores indicate better health outcomes.
Sleep Quality Assessment via Pittsburgh Sleep Quality Index (PSQI) | Baseline and 3 months
  Changes in sleep quality will be assessed using the PSQI questionnaire, which evaluates sleep quality over the past month. The PSQI produces a global score ranging from 0 to 21, with higher scores indicating worse sleep quality

OTHER OUTCOMES:
Anti-inflammatory effects of TRE | Baseline and 3 months
  Hypothesis-generating exploration and measure of anti-inflammatory effects of TRE assessed by plasma inflammatory cytokine levels.
Time in Range | Baseline and 3 months
  Change in the time spent within the target glucose range, as assessed by Continuous Glucose Monitoring (CGM) from interstitial glucose.
Glycemic Variability | Baseline and 3 months
  Change in glycemic variability, as assessed by Continuous Glucose Monitoring (CGM) from interstitial glucose.
Mean Glucose | Baseline and 3 months
  Change in mean glucose levels, as assessed by Continuous Glucose Monitoring (CGM) from interstitial glucose.

CONTACTS AND LOCATIONS:
Overall Officials: Pam Taub, MD, Principal Investigator — University of California, San Diego Health
Locations (1):
- Altman Clinical and Translational Research Institute, La Jolla, California, United States